CLINICAL TRIAL: NCT06734858
Title: A Multicenter, Randomized, Open-label, Controlled, Pivotal Clinical Trial to Evaluate the Efficacy and Safety of Software SAT-014 for the Alleviation of Symptoms Related to Trauma and Stressor-related Disorders
Brief Title: Pivotal Trial of SAT-014 for Trauma and Stressor-Related Disorder Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S-Alpha Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAT014-KP-002
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2024-12

CONDITIONS: Post-traumatic Stress Disorder; Adjustment Disorders
Keywords: post-traumatic stress disorder (PTSD); adjustment disorder (AD); SaMD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Adjustment Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAT014 study group (Experimental): SAT-0014 + Conventional treatment*
  *Conventional treatment: Pharmacological treatment received at baseline for the indication or simple counseling (excluding cognitive behavioral therapy and psychoanalytic counseling therapy)
  Interventions: Device: SAT014
- Control group (Other): Conventional treatment*
  *Conventional treatment: Pharmacological treatment received at baseline for the indication or simple counseling (excluding cognitive behavioral therapy and psychoanalytic counseling therapy)
  Interventions: Other: Control

INTERVENTIONS:
Device: SAT014 — SAT-014 in Combination with Baseline Conventional Treatment Participants in this arm will use the SAT-014 application for 6 weeks in combination with their baseline conventional treatment, which may include pharmacological therapy or simple counseling (excluding cognitive behavioral therapy and psychoanalytic counseling therapy). The aim of this study is to assess the efficacy and safety of SAT-014 for alleviating symptoms of trauma and stressor-related disorders, such as PTSD and adjustment disorder.
  Arms: SAT014 study group
Other: Control — Baseline Conventional Treatment Participants in this arm will receive only conventional treatment, which includes the medication they were taking at baseline for the indication or the basic counseling therapy they were receiving at baseline.
  Arms: Control group

SUMMARY:
The aim of this study is to evaluate the efficacy of SAt-014, a software as a medical device (SaMD), in alleviating symptoms of trauma and stressor-related disorders in patients with post-traumatic stress disorder (PTSD) or adjustment disorder (AD), compared to standard treatment, and to assess its safety for regulatory approval by the Ministry of Food and Drug Safety (MFDS).

DETAILED DESCRIPTION:
Stress-related mental disorders, including Post-Traumatic Stress Disorder (PTSD) and Adjustment Disorder (AD), are caused by traumatic experiences or significant stressors. These conditions can lead to social dysfunction, decreased quality of life, and increased suicide risk if untreated. With high global prevalence and rising patient numbers, existing treatments such as psychotherapy and pharmacotherapy have limitations. Digital therapeutics (DTx) offer a more accessible, cost-effective solution with less external exposure. Based on studies showing the effectiveness of therapies like EMDR and MBCT, SAT-014, a cognitive therapy software, was developed. An exploratory clinical trial was conducted to assess its initial safety and efficacy for alleviating symptoms of PTSD and AD. This trial, involving 110 participants over 19 years old, aims to evaluate SAT-014's efficacy in comparison with conventional treatments and assess its safety. The primary efficacy endpoint is the change in PCL-5 score at Week 6 (Visit 7) compared to baseline, while secondary endpoints include changes in PCL-5, IES-R, BAI, PHQ-9, HAM-A, CGI, and SF-12 scores at various time points.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years or older
* Diagnosed with Post-Traumatic Stress Disorder (PTSD) or Adjustment Disorder (AD) according to the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5)
* A score of 3 to 4 on the Clinical Global Impression-Severity (CGI-S) scale
* Able to access the internet and respond to app activity instructions
* Voluntarily decided to participate in this clinical trial and provided written consent by signing the participant information sheet and consent form

Exclusion Criteria:

* Those diagnosed with schizophrenia, bipolar disorder type 1, or psychotic disorders
* Those diagnosed with neurodevelopmental disorders, neurocognitive disorders, or organic mental disorders
* Those with severe depression (Patient Health Questionnaire-9 (PHQ-9) ≥ 20)
* Those with severe personality disorders
* Those diagnosed with substance use disorders (excluding nicotine and caffeine) or severe alcohol use disordes
* Those exhibiting active suicidal tendencies (suicidal thoughts, suicide attempts, or suicidal behavior)
* Those who have had a change in the type, dosage, or regimen of anxiolytics or antidepressants within 4 weeks of baseline
* Those currently participating in another clinical trial or who have participated in a clinical trial within 90 days prior to the screening visit
* Those deemed unsuitable for participation in the trial at the discretion of the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
Change in Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) score | baseline, 6 weeks
  The PTSD Checklist for DSM-5 (PCL-5) consist of 20 items, with a scale ranging from 0 to 4. Each item evaluates the frequency or intensity of specific symptoms over the past month. The scores are summed to produce a total severity score that ranges from 0 (minimum score) to 80 (maximum score). A higher scores indicate greater distress due to symptoms to past stressful experiences and a worse outcome.

SECONDARY OUTCOMES:
Change in Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) score | Baseline, 2 weeks, 4 weeks, 6 weeks
  PCL-5 consists of 20 items, with a scale ranging from 0 to 4. The scores range from 0 to 80, with higher scores indicating greater frequency and severity of PTSD symptoms.
Change in Beck Anxiety Inventory (BAI) score | Baseline, 2 weeks, 4 weeks, 6 weeks
  The Beck Anxiety Inventory (BAI) consists of 21 items, each assessing the intensity of anxiety symptoms experienced over the past week. Each item is rated on a 4-point scale, ranging from 0 (not at all) to 3 (severely-I could barely stand it). The total score can range from 0 to 63. Scores between 0 and 7 indicate minimal anxiety, while scores from 8 to 15 reflect mild anxiety. A score between 16 and 25 suggests moderate anxiety, and scores from 26 to 63 indicate severe anxiety. A higher score correlates with more severe anxiety.
Change in (Patient Health Questionnaire-9 (PHQ-9) score | Baseline, 2 weeks, 4 weeks, 6 weeks
  Change in PHQ-9 (Patient Health Questionnaire-9) score at each time point compared to baseline.
  The PHQ-9 (Patient Health Questionnaire-9) consists of 9 questions. Each question is scored on a 4-point scale, ranging from 0 (not at all) to 3 (nearly every day), resulting in a total score ranging from 0 to 27. The PHQ-9 score quantitatively reflects the severity of depressive symptoms, with higher scores indicating more severe depression.
Change in Hamilton Anxiety Scale (HAM-A) score | Baseline, 2 weeks, 4 weeks, 6 weeks
  The HAM-A (Hamilton Anxiety Rating Scale) consists of 14 items, with each item scored on a scale from 0 (not present) to 4 (extremely severe). The total score can range from 0 to 56. The HAM-A score reflects the severity of a patient's anxiety symptoms, with higher scores indicating more severe anxiety.
Change in Clinical Global Impression-Severity (CGI-S) score | Baseline, 2 weeks, 4 weeks, 6 weeks
  The CGI-S scale ranges from 1 to 7, with each score representing a different level of illness. Higher scores reflect more serious illness.
Clinical Global Impression-Improvement (CGI-I) score | Baseline, 2 weeks, 4 weeks, 6 weeks
  The CGI-I scale uses a 7-point rating system to assess improvement in a patient's condition.
  The CGI-I score ranges from 1 point (very much improved) to 7 points (very much worse). A higher score indicates that the symptoms have worsened.
Change in Impact of Event Scale - Revised (IES-R) score | Baseline, 2 weeks, 4 weeks, 6 weeks
  The Impact of Event Scale - Revised (IES-R) consists of 22 items, with each item rated on a 5-point scale, ranging from 0 (not at all) to 4 (extremely). The total score can range from 0 to 88. The IES-R total score reflects the severity of PTSD symptoms, with higher scores indicating a greater level of psychological distress and more intense post-traumatic stress responses.
Percentage of participants with a ≥10 point reduction in PTSD Checklist for DSM-5 (PCL-5) score | Baseline, 6 weeks
  The percentage of participants showing a greater than or equal to a 10-point reduction in their PTSD Checklist for DSM-5 (PCL-5) score will be measured at Week 6 (Visit 7) compared to baseline. PCL-5 consists of 20 items, each rated on a scale from 0 to 4. The total score ranges from 0 to 80, with higher scores indicating a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Hong, MD, Principal Investigator — Samsumg Medical Center; Kang, MD, Principal Investigator — Severance Hospital; Seo, MD, Principal Investigator — Wonju Severance Christian Hospital; Lee, MD, Principal Investigator — Kyung Hee University Hospital; Yoo, MD, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (5):
- South Korea (5):
  - Kyung Hee University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: No